CLINICAL TRIAL: NCT00908934
Title: An Open-label, Randomized, 2 Cohort, 2 Period Crossover Study to Assess the Relative Bioavailability of the Phase III to the Phase IIb Formulation of AZD9056 in Healthy Male and Female Subjects
Brief Title: AZD9056 Relative Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D1520C00004; EudraCT Number: 2009-010554-35
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: Relative Bioavailability; AZD9056

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 50 or 400 mg AZD9056, Test formulation
  Interventions: Drug: AZD9056 formulation Phase III 50 mg (T); Drug: AZD9056 formulation Phase III 200 mg (T)
- 2 (Experimental): 50 or 400 mg AZD9056, Reference formulation
  Interventions: Drug: AZD9056 formulation Phase IIb 50 mg (R); Drug: AZD9056 formulation Phase IIb 200mg (R)

INTERVENTIONS:
Drug: AZD9056 formulation Phase III 50 mg (T) — Given as 50 mg tablet (T)
  Arms: 1
Drug: AZD9056 formulation Phase IIb 50 mg (R) — Given as 50 mg tablet (R)
  Arms: 2
Drug: AZD9056 formulation Phase III 200 mg (T) — Given as 400 mg (2 x 200 mg tablet (T))
  Arms: 1
Drug: AZD9056 formulation Phase IIb 200mg (R) — Given as 400 mg (2 x 200 mg tablet (R))
  Arms: 2

SUMMARY:
The aims of this study are to compare the blood levels achieved with a new formulation of AZD9056 to an existing formulation of AZD9056 used in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures
* Healthy Volunteers, Females should not be of childbearing potential
* BMI between 18 and 30 kg/m2

Exclusion Criteria:

* Clinically significant ECG abnormality suggestive of underlying cardiovascular disease
* A history or presence of GI, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism and excretion of drugs
* Known or suspected drug or alcohol abuse or positive DOA test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-05; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of AZD9056 using PK variables Cmax and AUC | For each study period, intensive sampling occasions on day 1: half hourly after dosing until 4 hours, then 4,6,8 and 12 hours post dose, with once daily sampling on days 2 to 7

SECONDARY OUTCOMES:
Descriptive PK parameters for AZD9056 using PK variables (tmax, AUC(0-t), t1/2, CL/F and Vz/F) | For each study period, intensive sampling occasions on day 1: half hourly after dosing until 4 hours, then 4,6,8 and 12 hours post dose, with once daily sampling on days 2 to 7
Safety variables (adverse events, safety lab, blood pressure, pulse, ECG) | Frequent sampling occasions throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, Study Director — AstraZeneca R&D, Alderley Park, UK; Simon Constable, Principal Investigator — ICON Development Solutions, Manchester, UK
Locations (1):
- Research Site, Manchester, United Kingdom